CLINICAL TRIAL: NCT04477928
Title: Sanford Population Level Estimation of Type 1 Diabetes Risk GEnes in Children
Brief Title: General Population Level Estimation for Type 1 Diabetes Risk in Children During Routine Care Delivery
Acronym: PLEDGE
Status: Recruiting | Type: Observational
Sponsor: Sanford Health (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Pacific Northwest Research Institute (Other); University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: PLEDGE
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes; Celiac Disease
Keywords: Population screening; Type 1 Diabetes; Celiac Disease; Autoantibodies; Prevention; Diabetic Ketoacidosis (DKA); Genetic Risk Score; Differential Gene Expression; Economic Modeling; Quality of Life; Feasibility; Pragmatic; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Celiac Disease; Diabetic Ketoacidosis; Genetic Risk Score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Children receiving routine care at a Sanford facility
  Interventions: Diagnostic Test: Sera and whole blood sampling; Diagnostic Test: Differential Gene Expression (DGE)

INTERVENTIONS:
Diagnostic Test: Sera and whole blood sampling — * Study Entry: Single Nucleotide Polymorphism (SNP)-Based Genetic Risk Score at study entry.
  * 2 years old: T1D autoantibodies, Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) antibodies
  * 5 years old: T1D and celiac autoantibodies
  * 9-16 year old: one-time T1D and celiac autoantibodies
  * Siblings of people with T1D autoimmunity, ages 6-17 years: one-time T1D and celiac autoantibodies
Diagnostic Test: Differential Gene Expression (DGE) — Opt-in: Differential Gene Expression from cord blood at birth and peripheral blood at 12 months of age

SUMMARY:
In partnership with Helmsley Charitable Trust, the Sanford PLEDGE Study is a large-scale, observational, feasibility study of general population screening for T1D and celiac autoantibodies. Screening is incorporated into routine health care visits within an integrated health system.

DETAILED DESCRIPTION:
Most children with type 1 diabetes (T1D) do not have a family member with diabetes and often are not diagnosed until the child is very sick. Research suggests that screening and identifying children at risk for T1D autoantibodies can prevent serious illness at the time of diagnosis and improve long-term health outcomes.

The investigators will screen children, ages 0-5.99 or 9-16 years for blood markers related to T1D and celiac disease during routine healthcare delivery at birth, 1, 2 and 5 years, or once between 9 and 16 years of age. Children with confirmed autoantibodies will be offered participation in other monitoring or prevention trials (T1D), or referred to clinical care (celiac).

ELIGIBILITY:
Inclusion Criteria:

* Newborn Entry: Viable, term infants, defined as 36 weeks gestation by either dates or ultrasound who are born to pregnant women, 18 years or older, who are willing and able to provide informed consent (IC) prior to the onset of active labor. Who are born at a Sanford Health Hospital and plan to have routine well-child care at a Sanford Clinic
* Pediatric Entry: Children less than 6 years of age who receive their routine care at a Sanford facility and whose parents are able to provide IC.
* Adolescent Entry: Children, ages 9-16 years old, who receive their routine care at a Sanford facility and whose parents are able to provide IC.
* Siblings of children known to have T1D-relevant antibodies; ages 6 to 17 years old who receive care at a Sanford clinic
* Have an active MyChart account (with proxy access).

Exclusion Criteria:

* Subject is in the opinion of the investigator, unable to comply with the requirements of the study protocol.
* Children known to have T1D

Ages: 0 Minutes to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born at and/or followed at Sanford Health System facilities:
  1. . 0-5 years of age;
  2. . 9-16 years of age;
  3. . Siblings of children known to have T1D-relevant antibodies, ages 6 to 17 years old.
Sampling Method: Non-Probability Sample
Enrollment: 33000 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Demonstrated feasibility of large-scale population screening, as evidenced by: | By year 10 of the study
  1. The percentage of parent(s) that viewed the MyChart study information who went on to complete the MyChart informed consent, HIPAA and questionnaires.
  2. Of those who consented to be in the study, the percentage who went on to obtain the initial sample.
  3. Of the total samples collected, percentage that were valid and results received.
  4. The percentage of subjects who complete their ~60 month visit by their 6th birthday.

SECONDARY OUTCOMES:
Seroconversion rates for T1D-relevant and celiac autoantibodies | By year 10 of study
Percentage of T1D seropositive subjects who enroll in another T1D monitoring or prevention study. | By year 10 of study
Percentage of celiac seropositive subjects referred on to GI or primary care | By year 10 of study
The percentage of celiac seropositive subjects who were evaluated in clinical setting | By year 10 of study
The rate of development of overt hyperglycemia consistent with T1D (Stage 3). | By year 10 of study
Proportion of participants developing overt hyperglycemia consistent with T1D (Stage 3), who present in diabetic ketoacidosis (DKA) | By year 10 of study
Number and type of procedure-related adverse events | By year 10 of study
Assessment of costs associated with implementation of study compared to potential impacts on cost and quality of life. | By year 10 of study

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Griffin, PhD, MD, Principal Investigator — Sanford Research
Locations (4):
- United States (4):
  - Sanford Bemidji Region Clinics, Bemidji, Minnesota
  - Sanford Bismarck Region Clinics, Bismarck, North Dakota
  - Sanford Fargo Region Clinics, Fargo, North Dakota
  - Sanford Sioux Falls Region Clinics, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient characteristics, clinical and laboratory outcomes will be shared in an online platform.
Supporting Information: ICF, CSR
Time Frame: Data will be available no later than 12 months after the conclusion of study.
Access Criteria: Data available to researchers approved by investigators.

REFERENCES:
- [Background] Sims EK, Besser REJ, Dayan C, Geno Rasmussen C, Greenbaum C, Griffin KJ, Hagopian W, Knip M, Long AE, Martin F, Mathieu C, Rewers M, Steck AK, Wentworth JM, Rich SS, Kordonouri O, Ziegler AG, Herold KC; NIDDK Type 1 Diabetes TrialNet Study Group. Screening for Type 1 Diabetes in the General Population: A Status Report and Perspective. Diabetes. 2022 Apr 1;71(4):610-623. doi: 10.2337/dbi20-0054. PMID 35316839